CLINICAL TRIAL: NCT01034501
Title: Efficacy of Adjunctive Photodynamic Therapy in Non-surgical Treatment of Chronic Periodontitis: a Randomized , Controlled Clinical Trial
Brief Title: Adjunctive Photodynamic Therapy in Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Giorgio De Micheli, Associated, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP2112008
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Periodontitis
Keywords: periodontitis; photodynamic therapy
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- photodynamic therapy (Active Comparator): photodynamic therapy 660 nm,40 mW,60 Hz
  Interventions: Device: photodynamic therapy
- sham procedure (Sham Comparator): Not activation of laser device
  Interventions: Device: sham procedure

INTERVENTIONS:
Device: sham procedure — non activated laser tip
  Other Names: Laser Hand - MM Optics (ANVISA: 80051420009)
  Arms: sham procedure
Device: photodynamic therapy — photodynamic therapy 660 nm,40 mW,60 Hz
  Other Names: Laser Hand - MM Optics (ANVISA: 80051420009)
  Arms: photodynamic therapy

SUMMARY:
The aim of this study is to verify the efficacy of Photodynamic Therapy (PDT) as an adjunct to non-surgical treatment of chronic periodontitis by assessing clinical and microbiological and immunological parameters. This is a randomized, controlled, double-blind, parallel clinical trial. Thirty eight patients with chronic periodontitis will receive conventional periodontal treatment. After eight weeks, patients will be re-evaluated and sites with residual pockets (PD ≥ 5 mm ) will be selected as experimental sites, and will be allocated to test and control group randomly. The test group will receive the application of PDT and the control group will receive sham procedure. The clinical parameters will be evaluated at baseline, 3, 6 and 12 months after treatment. Subgingival plaque will be collected before PDT, a week after, 3, 6 and 12 months later. The microbiological evaluation will detect and quantify periodontal pathogens such as Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola and Aggregatibacter actinomycetencomitans with real time-PCR. During follow-up, patients will receive periodontal maintenance every 3 months, as well as the application of PDT or sham

DETAILED DESCRIPTION:
The goal of periodontal treatment is to restore tissue health through the elimination and control of etiologic factors, reducing the microbial aggression. Some microorganisms persist in the root surface even after scraping. Thus, the conventional mechanical treatment may fail to reduce the number of periodontal pathogens to levels compatible with health. This study will verify the efficacy of Photodynamic Therapy (PDT) as an adjunct to non-surgical treatment of chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Periodontitis (Tonetti, Claffey, 2005)
* 10 or more teeth
* 2 or more site with probing pocket depth ≥ 5 mm, with or without bleeding on probing, after re-evaluation

Exclusion Criteria:

* Profilatic antibiotics
* Diabetes, immunosuppression, pregnancy nursing mother
* Smoking
* Medication that might interfere with periodontal healing
* Previous periodontal treatment or antibiotics (6 months)
* Experimental teeth with mobility II or III, or endodontic problem

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in mean attachment level | 12 months

SECONDARY OUTCOMES:
Change in probing pocket depth | 12 months
Change in periodontal pathogens(Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola and Aggregatibacter actinomycetencomitans)counts. | 12 months
Change in fluid inflammatory markers (Il-1B, Il-6, Il-8, PGE2, TNF-a, Il-10, MMP-2, TIMP-1, MMP-8) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio De Micheli, Professor, Principal Investigator — FOUSP
Locations (1):
- Faculdade de Odontologia da Universidade de São Paulo (FOUSP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Christodoulides N, Nikolidakis D, Chondros P, Becker J, Schwarz F, Rossler R, Sculean A. Photodynamic therapy as an adjunct to non-surgical periodontal treatment: a randomized, controlled clinical trial. J Periodontol. 2008 Sep;79(9):1638-44. doi: 10.1902/jop.2008.070652. PMID 18771363
- [Background] Braun A, Dehn C, Krause F, Jepsen S. Short-term clinical effects of adjunctive antimicrobial photodynamic therapy in periodontal treatment: a randomized clinical trial. J Clin Periodontol. 2008 Oct;35(10):877-84. doi: 10.1111/j.1600-051X.2008.01303.x. Epub 2008 Aug 17. PMID 18713259
- [Derived] Carvalho VF, Andrade PV, Rodrigues MF, Hirata MH, Hirata RD, Pannuti CM, De Micheli G, Conde MC. Antimicrobial photodynamic effect to treat residual pockets in periodontal patients: a randomized controlled clinical trial. J Clin Periodontol. 2015 May;42(5):440-7. doi: 10.1111/jcpe.12393. Epub 2015 Apr 22. PMID 25808980